CLINICAL TRIAL: NCT04723836
Title: Optimal Nutrition for Prevention of Hypertension in Pregnancy Using a Personalised Approach
Brief Title: Optimal Nutrition for Prevention of Hypertension in Pregnancy
Acronym: OptiPREG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: DSM Ltd (Industry); Public Health Agency (Northern Ireland) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16/NI/0029
Record Dates: First submitted 2021-01-12; First posted 2021-01-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Blood Pressure; Pregnancy
Keywords: Pregnancy; Maternal blood pressure; MTHFR 677TT genotype; Riboflavin; 5-methyltetrahydrofolate; Offspring blood pressure
MeSH Terms: interventions — Riboflavin; 5-methyltetrahydrofolate

STUDY DESIGN:
Intervention Model Description: A double-blind randomised controlled trial embedded in a large longitudinal observational study in pregnant women.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- TT genotype active comparator group (Active Comparator): 5mg riboflavin per day from 16th gestational week
  Interventions: Dietary Supplement: Riboflavin (5mg)
- TT genotype experimental group (Experimental): 5mg riboflavin + 400µg 5-methyltetrahydrofolate per day from 16th gestational week
  Interventions: Dietary Supplement: Riboflavin (5mg); Dietary Supplement: 5-methyltetrahydrofolate (400µg)
- TT genotype placebo group (Placebo Comparator): Placebo supplement from 16th gestational week
  Interventions: Dietary Supplement: Placebo
- CT genotype active comparator group (Active Comparator): 5mg riboflavin per day from 16th gestational week
  Interventions: Dietary Supplement: Riboflavin (5mg)
- CT genotype experimental group (Experimental): 5mg riboflavin + 400µg 5-methyltetrahydrofolate per day from 16th gestational week
  Interventions: Dietary Supplement: Riboflavin (5mg); Dietary Supplement: 5-methyltetrahydrofolate (400µg)
- CT genotype placebo group (Placebo Comparator): Placebo supplement from 16th gestational week
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Riboflavin (5mg) — From 16th week gestation until end of pregnancy
  Other Names: Vitamin B2
  Arms: CT genotype active comparator group; CT genotype experimental group; TT genotype active comparator group; TT genotype experimental group
Dietary Supplement: 5-methyltetrahydrofolate (400µg) — From 16th week gestation until end of pregnancy
  Arms: CT genotype experimental group; TT genotype experimental group
Dietary Supplement: Placebo — From 16th week gestation until end of pregnancy
  Arms: CT genotype placebo group; TT genotype placebo group

SUMMARY:
The aim of this study is to investigate the role of the 677C→T polymorphism in the methylenetetrahydrofolate reductase (MTHFR) gene on blood pressure (BP) during pregnancy, and to examine the effect of intervention with riboflavin, alone or in combination with 5-methyltetrahydrofolate (5-MTHF), as a non-drug approach for managing BP in pregnancy in women with the variant TT genotype. In addition, we aim to examine the effect of maternal supplementation with riboflavin, alone or combined with 5-MTHF, on BP in the offspring in early infancy.

Study design: A double-blind randomized controlled trial embedded in a large longitudinal observational study in pregnant women will be conducted. Women with a singleton pregnancy who are in their first trimester will be recruited from antenatal clinics in Northern Ireland and the Republic of Ireland. Women interested in the study will provide informed consent, complete a screening questionnaire and will provide a buccal swab to collect DNA to screen for the MTHFR 677C→T polymorphism. Women with multiple pregnancies, a previous NTD-affected pregnancy and those who are taking medication interfering with B-vitamin metabolism will be excluded from participation in the study. At approximately the 16th gestational week (GW), those with the variant TT genotype and age-matched heterozygous women (CT genotype) will be randomised to receive riboflavin (5 mg/day) alone, or in combination with 5-MTHF (400µg/day), or placebo, until the end of pregnancy. A non-fasting blood sample will be collected for biomarker assessment of B-vitamin status and other relevant variables from each participant before intervention and at the 36th GW. At the same time points, anthropometric and BP measurements will be taken. Women will also complete a health and lifestyle questionnaire and a 4-day dietary record. Samples of cord blood, umbilical cord and placenta will be collected after delivery and anthropometric parameters of the newborns will be retrieved postpartum. Maternal and infant BP will be measured 2-4 and 36 months after birth. In parallel with the intervention trial, age-matched pregnant women who do not carry the variant gene (CC genotype) and have not been randomized to treatment, will be monitored in order to control for any changes associated with normal pregnancy in the study outcome measurements. In the pilot phase, the feasibility and acceptability of the study procedures and treatment will be evaluated for clarification of the sample size and refinement of the study protocol.

DETAILED DESCRIPTION:
The overall aim of this study is to investigate the role of a common genetic polymorphism in folate metabolism, MTHFR 677C→T, on blood pressure (BP) during pregnancy and the impact of B-vitamin supplementation as a non-drug approach for the management of BP in pregnancy in women with variant TT genotype.

Primary aims

1. To investigate BP in relation to MTHFR 677C→T polymorphism in pregnancy;
2. To investigate the response of BP during pregnancy to supplementation with riboflavin (5mg/d) alone, or in combination with 5-MTHF (400μg/d), targeted at women with the TT genotype;

Hypotheses:

* BP will be higher in women with the TT genotype compared to those with CT and CC genotype;
* Targeted supplementation with riboflavin during pregnancy will prevent the greater increase in BP observed in TT women compared to women with CC or CT genotypes;
* Supplementation with riboflavin in combination with 5-MTHF maybe more effective in preventing the greater increase in BP observed in TT women compared to women with CC or CT genotypes;

Secondary aims

1. To examine the effect of maternal supplementation with riboflavin (5mg/d) alone, or in combination with 5-MTHF (400μg/d), on BP of the offspring at 2-4 months and 3 years after birth in relation to this polymorphism;
2. To examine the relationship of riboflavin with haematological status and risk of anaemia
3. To examine the effect of riboflavin supplementation on change in haemoglobin concentrations
4. To evaluate the feasibility and acceptability of the study procedures to inform for the required sample size and refinements of the study protocol (pilot phase).

Hypotheses:

* Maternal supplementation with riboflavin, alone or riboflavin in combination with 5-MTHF, will influence the BP of newborns with TT genotype. In non-supplemented mothers, newborns with the TT genotype will have higher BP compared to newborns with CC and CT genotype. In supplemented mothers no genotype differences in newborns will be observed.
* Women with deficient biomarker status of riboflavin will have poorer haematological status and will be at greater risk of developing anaemia during pregnancy.
* Intervention with riboflavin will lead to improved haemoglobin concentrations compared to placebo.

In advance of their first antenatal appointment, participants will receive a participant information sheet from their obstetrician and those who are interested in the study will be referred by the staff at antenatal clinics to the OptiPREG research team. At baseline, pregnant women will provide a signed informed consent. Women with a singleton pregnancy who are in their first trimester of pregnancy will be eligible to take part in the study. Exclusion criteria will be: a high-risk pregnancy; a previous neural tube defect (NTD)-affected pregnancy or being the first degree relative of a woman who had a pregnancy affected with an NTD, or are themselves a sufferer of an NTD; use of medication known to interfere with B vitamin metabolism (Chloramphenicol, Methotrexate, Metformin, Sulfasalazine, Phenobarbital, Phenytoin, Primidone, Triamterene, Barbiturates). Those women who are eligible to take part in the study will provide at baseline a buccal swab to collect DNA for MTHFR genotyping, a non-fasting blood sample, and will have BP measured, along with weight and height measurements and will complete a health and lifestyle questionnaire and a 4-day food diary.

At 16th gestational week (GW), women with the TT genotype will be matched for age and systolic BP to women with the CT and CC genotypes. Although the primary purpose of the OptiPREG trial is to examine the effect of riboflavin intervention on BP in women with the TT genotype, those with the CT genotype will be also randomised to intervention (in a parallel trial). The purpose of this arm of the trial (in the CT genotype group) will be to identify any potential foetuses with the TT genotype so that their BP, and the impact of maternal B vitamin intervention, can be investigated. Within each genotype group (TT and CT), women will be stratified by systolic BP and age and will be randomized to receive 5 mg/day riboflavin, alone or in combination with 5-MTHF at 400µg/day, or placebo, until the end of pregnancy. In order to encourage maximal compliance, participants will be contacted regularly and provided with supplements in blister packs every 6 weeks during the intervention, and will be asked to return the blister packs; the number of unused capsules will be recorded to monitor compliance.

A second appointment will be organised at approximately the 36th GW when participants will provide a second non-fasting blood sample, will have BP and weight measurements taken and will provide information regarding any changes in health status, lifestyle and medication usage.

Following delivery, cord blood sample will be collected; dimensions and the weight of placenta will be measured, and placenta samples will be collected, together with a small section of the umbilical cord. The weight and length of the newborn, as well as the type of delivery and any complications in late pregnancy and birth will be retrieved from the mothers records postpartum.

In parallel with the TT and CT women on intervention, age-matched pregnant women with the CC genotype (not on intervention) will be monitored at the same time points (8-15 GW; 36 GW) in order to control for any changes in BP and other study outcome measurements associated with normal pregnancy.

Mother-child pairs will be visited at home when the offspring are 2-4 and 36 months. Weight, length and BP of the infant will be measured, and a buccal swab will be taken for MTHFR genotyping. Maternal BP and weight will be measured and mothers will be asked to provide information on health and lifestyle, infant feeding practice and health status. Additionally, at the 3 year appointment, offspring neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

• Women with a singleton pregnancy who are in their first trimester of pregnancy

Exclusion Criteria:

* Patients who have a high risk pregnancy, a previous pregnancy with a neural tube defect (NTD) or are the first degree relative of a woman who had a pregnancy affected by NTD or are themselves a sufferer of an NTD
* Women who are taking medication known to interfere with B-vitamin metabolism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women only
Enrollment: 2250 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Blood Pressure | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Taken according to the clinical guidelines in pregnancy from the UK National Institute for Health and Care Excellence (NICE)

SECONDARY OUTCOMES:
Vitamin B12 status | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Measured by a microbiological L. Leichmannii assay; serum methylmalonic acid concentrations by Gas Chromatography-Mass Spectrometry
Plasma homocysteine | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Measured using a fluorescence polarization immunoassay
Riboflavin status | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Measured using the erythrocyte glutathione reductase activation coefficient
Vitamin B6 status | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Plasma pyridoxal phosphate concentrations measured by High Performance Liquid Chromatography
Folate status | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Measured by a microbiological L.casei assay
MTHFR C677T polymorphism (rs1801133) | 12-week gestation (mother) and 2-4 or 36 months postpartum (offspring)
  Genotype of mother and offspring determined by restriction enzyme typing Hinf1 digestion in DNA extracted from buccal swabs
Maternal blood pressure | 2-4 and 36 months postpartum
  Taken according to the clinical guidelines in pregnancy from the UK National Institute for Health and Care Excellence (NICE)
Offspring blood pressure | 2-4 and 36 months after birth
Offspring anthropometry | 2-4 and 36 months after birth
  Length (cm)
Offspring anthropometry | 2-4 and 36 months after birth
  Weight (kg)
Maternal anthropometry | At baseline, 36 gestational week (weight only), 2-4 months postpartum (weight only)
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2
Placenta size | At birth
  Placenta weight (g)
Placenta size | At birth
  Dimensions (cm)
Placenta and umbilical cord histology | At birth
  Samples will be examined for villous changes (i.e. presence of infarcts, increased syncytial knots and fibrin deposition, hyalinized avascular villi) and vascular lesions (i.e. decidual vascular thrombosis, spiral artery fibrinoid necrosis, mural hypertrophy of decidual arterioles, thrombi in large fetal vessels, fibromuscular sclerosis in intermediate-sized fetal vessels)
Offspring neurodevelopment | 36 months post birth
  Assessed by Bayley Scales of Infant and Toddler Development (0-19 across 5 domains). The higher the score the more progressed the child's development.
Haemoglobin concentration | Change between baseline (12th week gestation) and end of intervention (36 week gestation)
  Change in haemoglobin concentration as measured by SYSMEX analyser (g/L)
Presence of maternal anaemia | Change between baseline (12-week gestation) and end of intervention (36-week gestation)
  Defined as Hb <115g/L in the first and third trimesters or Hb<110 g/L in the second trimester

CONTACTS AND LOCATIONS:
Locations (3):
- Letterkenny University Hospital, Letterkenny, Ireland
- United Kingdom (2):
  - Northern Health and Social Care Trust, Coleraine, N.Ireland
  - Western Health and Social Care Trust, Londonderry, N.Ireland

IPD SHARING:
Plan to Share IPD: Undecided